CLINICAL TRIAL: NCT06937645
Title: the Effect of Hyaluronic Acid Platelets Rich Plasma on the Endometrial Receptivity and Intracytoplasmic Sperms Injection Outcome
Brief Title: the Effect of Hyaluronic Acid Intrauterine Wash on Endometrial Receptivity and Pregnancy Outcome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, ghada bassim raaf, clinical professor, Al-Nahrain University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0701-PF-2023G12
Record Dates: First submitted 2025-03-22; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Infertile Patients
Keywords: hyaluronic acid; intrauterine wash; endometrial receptivity; pregnancy outcome
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- the uterine cavity washed with hyaluronic acid preparation on the day of ooc (Experimental): 40 infertile patients had their uterine cavity with hyaluronic acid preparation on the day of oocytes retrieval in ICSI
  Interventions: Drug: Hyaluronic Acid (HA)
- 40 infertile females had their uterine cavity washed with PRP preparation (Experimental): 40 infertile females had their uterine cavity washed with PRP preparation on the day of oocytes retrieval in ICSI
  Interventions: Drug: platlet rich plasma (PRP)
- 40 infertile females with no intervention for their uterus (No Intervention): 40 infertile females with no intervention for their uterus on the day of oocytes retrieval in ICSI

INTERVENTIONS:
Drug: Hyaluronic Acid (HA) — hyaluronic acid PRP preparation used to wash the endometrium on the day of oocytes retrieval
  Arms: the uterine cavity washed with hyaluronic acid preparation on the day of ooc
Drug: platlet rich plasma (PRP) — PRP preparation used to wash the uterine cavity on the day of oocytes retrieval
  Arms: 40 infertile females had their uterine cavity washed with PRP preparation

SUMMARY:
Hyaluronic acid intrauterine wash is done for infertile females undergoing intracytoplasmic sperm injection on the day of oocyte retrieval. endometrial receptivity parameters, including the subendometrial vasculature indices were measured before and after the intervention for purpose of studying the effect of hyaluronic acid on improvement of the endometrial receptivity and subsequently the pregnancy outcome

ELIGIBILITY:
Inclusion Criteria:

* Infertile females aged 18-40 years.
* Infertile females scheduled for GnRH antagonist protocol of fresh ICSI cycle.
* Females use dual stimulation (GnRH agonist plus Ovetrelle) for ovulation triggering.

Exclusion Criteria:

* Infertile females diagnosed as a poor responder.
* Infertile females diagnosed with uterine pathology.
* Infertile females who are scheduled for a frozen ICSI cycle.
* Infertile females diagnosed with endocrine diseases like thyroid disease, diabetes mellitus, and hyperprolactinemia.
* Infertile females diagnosed with thrombocytopenia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
measuring the value of resistance index (RI) of the sub-endometrial blood vessels | for each participant twice measure will be done for (RI). The first measure will be performed on the day of oocyte retrieval and the second measure on the day of embryo transfer which is done 3-5 days after oocyte retrieval.
  We will measure the value of the resistance index (RI) using the transvaginal ultrasound Doppler study. For each patient, RI will be measured twice: the first measure will be done before the intervention on the day of oocyte retrieval, and the second measure will be performed after the intervention on the day of embryo transfer.
  we will calculate RI according to the following equation Resistance index (RI)= [Peak Systolic Velocity (PSV) cm/sec - End Diastolic Velocity (EDV) cm/sec ] / Peak Systolic Velocity (PSV) cm/sec Then a statistical comparison will be made to evaluate the difference between the two readings to study the effect of the intervention on the measured parameter for each group.
measuring the value of sub- endometrial vessels pulsatile index (PI) | for each participant twice measure will be done for PI. The first measure is on the day of oocyte retrieval and the second measure on the day of embryo transfer which is done 3-5 days after oocyte retrieval.
  We will measure the value of the pulsatile index (PI) using the transvaginal ultrasound Doppler study. PI will be measured twice for each patient: once before the oocyte retrieval intervention and once after the embryo transfer intervention.
  then PI will be calculated according to the following equation Pulsatility Index (PI) = [Peak Systolic Velocity (PSV) cm/sec - end Diastolic Velocity (EDV) cm/sec ] / Mean Velocity (MV) cm/sec Then a statistical comparison will be made to evaluate the difference between the two readings to study the effect of the intervention on the measured parameter for each group.
measuring the value of peak systolic to end diastolic ratio (S/D) of the sub-endometrial blood vessels | for each participant twice measure will be done for S/D. The first measure is on the day of oocyte retrieval and the second measure on the day of embryo transfer which is done 3-5 days after oocyte retrieval.
  We will measure the value of the peak systolic to end diastolic ratio (S/D) using the transvaginal ultrasound Doppler study. For each patient, S/D will be measured twice: the first measure will be done before the intervention on the day of oocyte retrieval, and the second measure will be performed after the intervention on the day of embryo transfer.
  S/D will be calculated according to the following equation S/D= Peak Systolic Velocity (PSV) cm/sec /End Diastolic Velocity (ED) cm/sec
  Then a statistical comparison will be made to evaluate the difference between the two readings to study the effect of the intervention on the measured parameter for each group.

SECONDARY OUTCOMES:
measuring serum level of beta human chorionic gonadotropin | 2 weeks from the day of oocyte retrieval
  We will assess the effect of hyaluronic acid intrauterine wash on improving the pregnancy outcome in infertile patients undergoing intracytoplasmic sperm injection (ICSI). Two weeks after the day of oocyte retrieval, we will measure the serum level of beta human chorionic gonadotropin (B HCG) in mIU/mL to test for successful pregnancy. The pregnancy rates will be compared between the study groups using statistical analysis to see how effective hyaluronic acid intrauterine wash is on pregnancy outcomes compared to the PRP and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- high institute for infertility diagnosis and ARTS, AL-Kadimya, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No